CLINICAL TRIAL: NCT06761105
Title: Observation of the Use of Digital Tools for Medical History-Taking in Primary Care and Utilization of Anonymous Routine Data for Health Services Research
Brief Title: Using Anonymous Data from a Digital Tool for Medical History-Taking to Improve Healthcare Services
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Goettingen (Other)
Responsible Party: Principal Investigator, Frank Müller, MD, PhD, MSc, MD PhD, University Hospital Goettingen
Other Study IDs: 4/8/24
Record Dates: First submitted 2024-12-05; First posted 2025-01-07 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-01

CONDITIONS: Health Services Research
Keywords: digital medical history; anonymized usage data; general practice; GP consultations; GP; health services research

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Patients who have used the digital medical history tool in one of the participating general practices

SUMMARY:
This study aims to understand how people use a mobile app that helps them record their symptoms before going to the doctor. Patients use the app on a tablet or other digital device. The app guides patients through a series of structured questions tailored to their symptoms. The data collected is then transferred to the practice's electronic record and is available to the treating doctor before and during the consultation.

In this project, anonymized usage data will be analyzed to contribute to the further development of the tool and to provide valuable insights for health services research.

DETAILED DESCRIPTION:
In several studies the usability of digital medical history tools has been demonstrated. These tools allow acute complaints to be recorded using an app before a medical consultation and the data collected to be transferred to the electronic medical record.

The aim of the study is to investigate the effectiveness and use of a digital medical history tool that is becoming increasingly popular in general practice. To this end, it is aimed to evaluate anonymized usage data provided by the company that distributes the app, aidminutes gUG, as part of an observational study with the aim of identifying potential for further development and for questions of health services research (e.g. on the frequency of GP consultations, morbidity and frequency of complaints). This is a retrospective data analysis of anonymous routine data in a cross-sectional design.

ELIGIBILITY:
Inclusion Criteria:

* all patients that use the app in a general practice that agreed to provide data
* all ages (including children if the app is used by parent or legal guardian)
* all complaints chosen in the app

Exclusion Criteria:

* patients that use the app in a general practice that did not agree to provide data
* patients that use the app in a general practice outside of the federal state Lower Saxony

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Lower Saxony, Germany
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2032-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Use patterns | From enrollment to the end of app use, up to 8 years
  Evaluation of the use patterns and frequencies of the medical history tool

SECONDARY OUTCOMES:
Data quality | From enrollment to the end of app use, up to 8 years
  Investigation of the consistency and completeness of the medical history data collected by the medical history tool

CONTACTS AND LOCATIONS:
Locations (1):
- Department of General Practice, Göttingen, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Needs to be discussed with responsible data officer